CLINICAL TRIAL: NCT02851420
Title: Interest of Spectroscopy in the Diagnosis of Cancerous and Precancerous Lesions of the Upper Airways (UA): Pilot Study
Brief Title: Spectrometry of Cancerous Lesions of the Oral Cavity
Acronym: SpectrORL1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FLAUS-BOZORG GRAYELI 2014
Record Dates: First submitted 2016-07-28; First posted 2016-08-01 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-09

CONDITIONS: Cancerous Lesions of the Oral Cavity
MeSH Terms: interventions — Spectrum Analysis

ARMS (2):
- control (Placebo Comparator)
  Interventions: Other: spectroscopy
- patient (Experimental)
  Interventions: Other: spectroscopy

INTERVENTIONS:
Other: spectroscopy

SUMMARY:
The detection of suspect lesions is based on the clinical examination of the oral cavity and pharyngolaryngeal endoscopy, but the examination to confirm the diagnosis is a pathology examination of the biopsy taken during the endoscopy. Taking the biopsy, however, can be difficult. On the one hand , it is an invasive procedure, and may engender complications, and on the other hand, certain modifications of the mucosa may be discrete, or not particularly specific or, on the contrary, disseminated or extremely widespread.

Non-invasive tools to help the diagnosis could prove to be particularly interesting 1) to restrict the use of biopsies to patients in whom it is really necessary 2) and to identify the area where the biopsy should be done in cases of multiple lesions. In this context, spectroscopy could be a promising alternative.

The investigator puts forward the hypothesis that cancerous and precancerous lesions of the mucosa of the upper airways and digestive tract present a characteristic spectrometric profile. Indeed, as malignant tumours are hypervascularized and as precancerous tumours show signs of angiogenesis, investigators expect that the reflectance of haemoglobin will be diminished in the specific wavelengths of 540 and 575 nm, corresponding to the principal wavelengths absorbed by haemoglobin.

This pilot study will make it possible to construct an algorithm that could be used to classify lesions of the upper airways and digestive tract as either seemingly benign or cancerous.

ELIGIBILITY:
Inclusion Criteria:

patient - Patients consulting at the oto rhino laryngology department of Dijon for a functional symptom of the mouth, pharynx or larynx (pharyngeal discomfort, odynophagia, dysphagia, dysphonia, laryngeal dyspnoea) and in whom the clinical examination reveals a suspect lesion of the oral cavity, the pharynx or larynx and imposes an endoscopy procedure under general anaesthesia (unless it is a lesion of the tonsils or lingual tonsils)

* Subjects who have provided consent
* Subjects over 18 years old

volunteers:- Volunteers

* Absence of risk factors cancerous oro-pharyngeal lesions, that is to say, non-smokers, alcohol consumption < 1 glass per day.
* Absence of functional oto rhino laryngology symptoms (dyspnoea, dysphagia, dysphonia, pain)
* Subjects who have provided consent
* Subjects over 18 years old

Exclusion Criteria:

patient :- Patients without national health insurance cover

* Pregnant or breast-feeding women
* Biopsies not feasible

  * because of difficulty of exposure of the tumour
  * tumour not accessible to the biopsy forceps,
  * complications during the procedure making it impossible to do the biopsies (difficulties with ventilation)
* Spectrometry not feasible

  * If exposure is difficult, tumour not accessible to the spectrometry probe (for example, a hypopharyngeal tumour in a patient with limited mouth opening)
  * In cases of anaesthesia complications, such as difficulties with ventilation
* Lesions of the tonsils or lingual tonsil, suggesting lymphoma (exclusion of lymphoid tumours)

volunteers:- Persons without national health insurance cover

* Pregnant or breast-feeding women
* Presence of risk factors: alcohol-smoking
* Presence of oto rhino laryngology functional symptoms

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2016-02-15 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2019-06-13 (Actual)

PRIMARY OUTCOMES:
Reflectance spectrum of haemoglobin | Day one

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Dijon Bourgogne, Dijon, France